CLINICAL TRIAL: NCT04747379
Title: Psychological Effect of Explicit Recall After Sedation
Brief Title: Psychological Effect of Explicit Recall After Sedation (PEERS)
Acronym: PEERS
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Jason Chui, Anesthesiologist/Associate Professor, Western University, Department of Anesthesia and Perioperative Medicine, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 114966
Record Dates: First submitted 2020-10-27; First posted 2021-02-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Awareness, Anesthesia; Post Traumatic Stress Disorder; Depression
Keywords: recall; awareness; sedation; post-traumatic stress disorder; trauma; depression; suicide; anesthesia
MeSH Terms: conditions — Intraoperative Awareness; Stress Disorders, Post-Traumatic; Depression; Wounds and Injuries; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Awareness, or explicit recall, under sedation is often intended and expected by anesthesiologists and is assumed that does not associate with any sequelae. Thus, awareness under sedation is a common event and is estimated to occur in around one-quarter of patients in our population. However, two recent studies suggested some patients with awareness under sedation have comparable psychological sequelae to those patients with awareness during general anesthesia. As such, we plan to conduct a a single center, prospective cohort study to determine the incidence of explicit recall under sedation/regional anaesthesia in adults, and to identify whether explicit recall experiences - or specific elements of those experiences (e.g. feeling pain and paralysis) - were associated with psychiatric sequelae.

In this study, we will prospectively include 2500 patients who will be scheduled to have total hip and knee joint replacement surgery under regional anesthesia and sedation at University Hospital, London Health Sciences Center.

All participants will be assessed at four separate time points including:

1. Enrollment/Surgical Preparatory Area (~ 2 hours before surgery)
2. Post Anesthesia Care Unit (assessment will be conducted in PACU prior to discharge, within a maximum window of 6 hours from PACU admission)
3. Postoperative day one (in hospital)
4. Postoperative 6 weeks (expected to be after discharge via telephone or in-person in clinic)

DETAILED DESCRIPTION:
Demographic and perioperative variables will be summarized. Descriptive statistics will be used to examine the incidence of awareness under sedation. We will further report the incidence of awareness with or without psychological sequalae, as well as the immediate and delayed awareness. We will also summarize the recall experience, initial emotional responses toward the event of awareness, as well as the patient satisfaction.

The psychological consequences will be defined and graded using the PHQ-9 (patient health questionnaire-9) and PCL-S (PTSD Checklist Stressor - S) questionnaires. The severity of harm using modiﬁed National Patient Safety Agency (NPSA) will also be described.

For the primary analysis, to assess the risk of explicit recall experience towards the development of PTSD and depression, we performed univariable logistic regression to assess whether explicit recall will be associated with either co-primary outcome. This will be followed by an assessment of individual element of recall experiences, such as auditory recall, feeling pressure, feeling pain and paralysis, etc. Multivariable logistic regression analysis will also performed to adjust for potential confounders

For the secondary analysis, we will further perform logistic regression analysis to assess the potential risk factors for explicit recall. The potential risk factors to fit into the models include: i) patient factors: obesity, obstructive sleep apnoea or any cardiopulmonary diseases that lead to sedation failure, history of psychiatric disease, ii) anestheteic factors such as the choice of sedatives, iii) patient expectation (assessed by NAP5 method), iv) duration and experiences of explicit recall (e.g. auditory, tactile or pain).

Additionally, we will assess patient expectations and communication between the patients and healthcare providers.

To assess the impact of surgery on the development of psychiatric symptoms, we will evaluate changes in the severity of depressive symptoms before and after surgery. We will also estimate the mental healthcare burden by determining the number of new psychiatric consultations potentially required.

P values <0.05 were accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (> or = 18 years old)
2. Scheduled to have orthopedic surgery or joint replacement therapy under sedation/regional anesthesia
3. Patient is able to communicate in English
4. ASA I-IV

Exclusion Criteria:

1. Unable to obtain informed consent
2. Patient received General Anesthesia (GA) or conversion to GA during their surgical procedures
3. Unable to conduct the survey such as language barrier, overt psychiatric disorder thought to interfere with the reliability of the interview (e.g. dementia etc)
4. Patient who is expected to require mechanical ventilation at postoperative period (i.e. unable to perform surveys at Post-Anesthesia Care Unit (PACU) and postoperative day one)
5. Unable to follow up via phone or attend a postoperative follow-up visit at postoperative 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo orthopedic or joint replacement surgeries under sedation/regional anesthesia at University Hospital located in London, Ontario, Canada.
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Explicit recall | Assessment will be conducted in PACU prior to discharge, within a maximum window of 6 hours from PACU admission
  Explicit recall will be assessed by Modified Brice Questionnaire

SECONDARY OUTCOMES:
Explicit Recall | Postoperative Day 1
  Explicit recall will be assessed by Modified Brice Questionnaire
  The Michigan Awareness Classiﬁcation is used to report the levels of sensation during awareness. 5 Levels of sensation are classiﬁed as auditory, tactile, pain, paralysis, or pain and paralysis. A designation of 'D' for distress is used for patient reports of fear, anxiety, suffocation, sense of doom, sense of impending death, or similar reports that indicated emotional distress during the explicit recall experience.
Sensation During Awareness | Postoperative Day 1
  The Michigan Awareness Classification - Michigan Score
  The Michigan Awareness Classiﬁcation is used to report the levels of sensation during awareness. 5 Levels of sensation are classiﬁed as auditory, tactile, pain, paralysis, or pain and paralysis. A designation of 'D' for distress is used for patient reports of fear, anxiety, suffocation, sense of doom, sense of impending death, or similar reports that indicated emotional distress during the explicit recall experience.
Details of recall experience | Postoperative Day 1
  Light, smell, and other feelings
  The Michigan Awareness Classiﬁcation is used to report the levels of sensation during awareness. 5 Levels of sensation are classiﬁed as auditory, tactile, pain, paralysis, or pain and paralysis. A designation of 'D' for distress is used for patient reports of fear, anxiety, suffocation, sense of doom, sense of impending death, or similar reports that indicated emotional distress during the explicit recall experience.
Post Traumatic Stress Disorder | Postoperative 6 weeks
  PCL-C Questionnaire
Depression | Postoperative 6 weeks
  PHQ-9 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, MD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- London Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided